CLINICAL TRIAL: NCT03530579
Title: Community Health Worker Diabetes Prevention Intervention
Acronym: RICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 11-01416
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Prevention
Keywords: Diabetes Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants will receive 6 two and a half hour educational group trainings over the course of 6 months.
  Interventions: Behavioral: Educational group trainings
- Group 2 (Active Comparator): A community health worker will answer your questions about diabetes and refer participant if you need one.
  Interventions: Behavioral: Community Health Care Worker

INTERVENTIONS:
Behavioral: Educational group trainings — Participants will receive 6 two and a half hour educational group training's over the course of 6 months. These sessions will be led by a trained CHW in your language and will be held on a monthly basis in a community based location.
  Session 1: What is Diabetes
  * Why is Prevention Important
  Session 2: Nutrition Session 3: Physical Activity Session 4: Cardiovascular Disease & Diabetes Complication Session 5: Stress Management Session 6: Access to Service
  Arms: Group 1
Behavioral: Community Health Care Worker — A community health care worker answer your questions about diabetes and refer participant to a physician. Survey will be completed at the start of the study and during the 3rd, 6th and 12th months
  Arms: Group 2

SUMMARY:
The primary goal of this study is to develop, implement, and test a community health worker (CHW) program designed to promote diabetes prevention among Korean and South Asian Americans in New York City.

In particular, the specific aims of this study are:

1. To utilize community based participatory research (CBPR) methods to expand upon an existing campus-community partnership to develop and implement a CHW program among Korean and South Asian Americans that promotes diabetes prevention;
2. To develop, implement, and assess the efficacy of a CHW intervention to promote diabetes prevention and access to care among NYC Koreans and South Asians.

ELIGIBILITY:
Inclusion Criteria:

* is a South Asian or Korean American immigrant;
* is identified as at-risk by a diabetes risk assessment
* is between 18-75 years of age; and
* is willing to be randomized to either treatment or control groups.

Exclusion Criteria:

* is a confirmed diabetic;
* is on renal dialysis;
* has an acute or terminal illness or serious mental illness;
* has a history of recent coronary event within the last 12 months;
* has a recent history of acute medical problem or admission to hospital;
* has any other severe medical conditions that might make it difficult to attend educational sessions;
* has poor short-term prognosis (expected death in <2 years);
* is planning to travel for longer than 6 weeks during the 6-month intervention period; or
* is participating in another CVD study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 954 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2015-02-13 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Change in weight | 3 Months, 6 Months, 12 Months
Change in Body Mass Index | 3 Months, 6 Months, 12 Months
Change in hip-to-waist ratio measurements | 3 Months, 6 Months, 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Islam, PhD, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wyatt LC, Katigbak C, Riley L, Zanowiak JM, Ursua R, Kwon SC, Trinh-Shevrin C, Islam NS. Promoting Physical Activity Among Immigrant Asian Americans: Results from Four Community Health Worker Studies. J Immigr Minor Health. 2023 Apr;25(2):291-305. doi: 10.1007/s10903-022-01411-y. Epub 2022 Oct 23. PMID 36273386